CLINICAL TRIAL: NCT04569305
Title: Principal Investigator
Brief Title: Effect of Negative Pressure Wound Therapy for Soft Tissue Injuries of Foot and Ankle in Patients at a Tertiary Care Hospital
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Roqayyah Munawwer Khursheed, Principal Investigator, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1408
Record Dates: First submitted 2020-09-18; First posted 2020-09-29 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Soft Tissue Injuries
MeSH Terms: conditions — Soft Tissue Injuries | interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Who Masked: Participant
Masking Description: This study will be single blinded means that patient will be unaware of his/her treatment method.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Negative Pressure Wound Therapy (Experimental): Negative Pressure Wound Therapy was applied to injured area of foot and ankle after debridement and cleaning of the necrosed/dead tissue. The effect of technique was assessed through measuring wound surface area covered with healthy granulation tissue measured in centimetre square on follow-up.
  Interventions: Procedure: Negative Pressure Wound Therapy
- Conventional treatment (Active Comparator): Simple moist gauze dressing applied to injured area of foot and ankle after debridement and cleaning of the necrosed/dead tissue. The effect of treatment was assessed through measuring wound surface area covered with healthy granulation tissue measured in centimetre square on follow-up.
  Interventions: Procedure: Conventional treatment

INTERVENTIONS:
Procedure: Negative Pressure Wound Therapy — NPWT technique was applied to injured area of the foot and ankle after debridement and cleaning of the necrosed tissue and using Vacuum Assisted Closure (VAC) consisting of evacuation tube, vacuum pump, collecting canister and a multiporous polyurethane sponge. VAC dressings were changed every 72 hours.
  Arms: Negative Pressure Wound Therapy
Procedure: Conventional treatment — In conventional treatment moist gauze dressings were applied and change of dressings were done daily.
  Arms: Conventional treatment

SUMMARY:
Effect of Negative Pressure Wound Therapy for Soft Tissue Iinjuries of Foot and Ankle in Patients at a Tertiary care Hospital.

To evaluate the effect of negative pressure wound therapy for soft tissue injuries of foot and ankle.This will be assessed through measuring the wound surface area covered with healthy granulation tissue measured in centimetre square on follow-up.

DETAILED DESCRIPTION:
All patients aged 18 years or above with foot and ankle trauma resulting in soft tissue injury with or without bones and tendon exposed were included in the study. 35 patients were randomized into Negative Pressure Wound Therapy group and 35 in conventional treatment group.In NPWT group ,NPWT was applied to injured area of foot and ankle after debridement and cleaning of the necrosed/dead tissue. The effect of technique was assessed through measuring wound surface area covered with healthy granulation tissue measured in centimetre square on follow-up at 10 days ,20 days and 27 days respectively.

In Conventional treatment group patients were kept on simple moist gauze dressings and the wound was assessed through measuring wound surface area covered with healthy granulation tissue measured in centimeter square on followup at 10 days , 20 days and 27 days respectively.

ELIGIBILITY:
Inclusion Criteria:

1. All patients aged 18 years or above with foot and ankle trauma resulting in soft tissue injury with bones and tendon exposed
2. Patients consenting to participate in the study

Exclusion Criteria:

1. Patients with uncontrolled diabetes mellitus
2. Patients with multiple fractures

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
size of wound covered with healthy granulation tissue | 27 days
  The effect of technique was assessed through measuring wound surface area covered with healthy granulation tissue measured in centimetre square on follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Roqayyah M Khursheed, MBBS, Principal Investigator — Dow University of Health Sciences
Locations (1):
- Roqayyah Munawwer Khursheed, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee HJ, Kim JW, Oh CW, Min WK, Shon OJ, Oh JK, Park BC, Ihn JC. Negative pressure wound therapy for soft tissue injuries around the foot and ankle. J Orthop Surg Res. 2009 May 9;4:14. doi: 10.1186/1749-799X-4-14. PMID 19426531
- See also: Negative pressure wound therapy for soft tissue injuries around the foot and ankle — http://www.josr-online.com/content/4/1/14